CLINICAL TRIAL: NCT01338883
Title: A Phase 2b Randomized, Double-Blind, Double-Dummy Trial of 100 or 200 mg Once-Daily Doses of Cenicriviroc (CVC, TBR 652) or Once-Daily EFV, Each With Open-Label FTC/TDF, in HIV 1-Infected, Antiretroviral Treatment-Naïve, Adult Patients With Only CCR5-Tropic Virus
Brief Title: Efficacy, Safety, and Tolerability of Cenicriviroc (CVC) in Combination With Truvada or Sustiva Plus Truvada in HIV 1-infected, Antiretroviral Treatment-naïve, Adult Patients Infected With Only CCR5-tropic Virus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tobira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TBR-652-2-202
Record Dates: First submitted 2011-04-18; First posted 2011-04-20 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: HIV-1 Infection
Keywords: HIV-1 Infection; CCR5-tropic; Anti-retroviral naive
MeSH Terms: interventions — cenicriviroc; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; efavirenz

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CVC 100 mg + Truvada (Experimental)
  Interventions: Drug: Cenicriviroc 100 mg
- CVC 200 mg + Truvada (Experimental)
  Interventions: Drug: Cenicriviroc 200 mg + Truvada
- Sustiva + Truvada (Active Comparator)
  Interventions: Drug: Sustiva + Truvada

INTERVENTIONS:
Drug: Cenicriviroc 100 mg — 100 mg CVC plus Truvada
  Arms: CVC 100 mg + Truvada
Drug: Cenicriviroc 200 mg + Truvada — 200 mg CVC plus Truvada
  Arms: CVC 200 mg + Truvada
Drug: Sustiva + Truvada — Sustiva plus Truvada
  Arms: Sustiva + Truvada

SUMMARY:
This is a randomized, double-blind, double-dummy, 48-week, comparative study. Approximately 150 HIV-infected, treatment-naïve patients with CCR5-tropic virus will be stratified by HIV-1 RNA: ≥100,000 copies/mL versus <100,000 copies/mL and will be randomized 2:2:1 to receive:

* Arm A: CVC 100 mg (2 tablets, 50 mg each) QD + CVC matching placebo (2 tablets) QD + EFV matching placebo (1 tablet) QHS + FTC/TDF (1 tablet) QD.
* Arm B: CVC 200 mg (4 tablets, 50 mg each) QD + EFV matching placebo (1 tablet) QHS + FTC/TDF (1 tablet) QD.
* Arm C: CVC matching placebo (4 tablets) QD + EFV 600 mg (1 tablet) QHS + FTC/TDF (1 tablet) QD.

Doses of both CVC/placebo and EFV/ placebo will be administered as double-blinded study drug. FTC/TDF will be administered as open-label study drug in a fixed-dose combination formulation (Truvada). CVC/placebo should be taken following breakfast; EFV should be taken on an empty stomach at bedtime.

HIV-1 RNA levels and CD4+ and CD8+ cell counts, percentages, and ratios will be measured at every visit. Samples for viral tropism and resistance testing in case of virologic failure will be collected at Screening and each on-treatment visit.

Biomarkers associated with inflammation and immune activation will be measured at Baseline (predose) and each study visit thereafter, with flow cytometry obtained at weeks 4, 12, 24, 48, and 52.

Fasting metabolic indicators of glucose control (glucose and insulin for HOMA-IR, HbA1c) and fasting lipid profiles (HDL, LDL, total cholesterol, and triglycerides) will be measured at Baseline (predose) and Weeks 4, 12, 24, 48, and 52. Waist-to-hip ratios will be measured at Baseline and Weeks 24 and 48.

Plasma samples will be collected and stored for possible future studies at Baseline (predose) and every visit thereafter.

ELIGIBILITY:
Selected Inclusion Criteria:

1. Adult male and female, HIV-1-infected patients 18 years old and older.
2. Body mass index (BMI) 18 to < 35 kg/m2.
3. Antiretroviral treatment-naïve. Treatment-naïve is defined as:

   * No prior nonnucleoside reverse transcriptase inhibitor, other than in women who received a single dose of perinatal nevirapine who have no K103 viral mutation.
   * No prior CCR5 antagonist therapy.
   * No more than 10 days of any other prior antiretroviral therapy.
4. HIV-1 CCR5-tropic-only virus.
5. Plasma HIV-1 RNA level >/=1,000 copies/mL at first Screening.
6. CD4 cell count >/=250 cells/mm3 at first Screening.

Selected Exclusion Criteria:

1. Presence of CXCR4- or dual/mixed-tropic HIV-1 virus.
2. Presence of primary resistance mutations or phenotypic resistance to TDF, FTC, or EFV and/or mutations associated with multidrug nucleoside/nucleotide resistance.
3. An active CDC category C disease (except cutaneous Kaposi's sarcoma not requiring systemic therapy during the trial).
4. Any historical CD4 count < 200 cells/mm3.
5. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value Grade > 2 or total bilirubin greater than the upper limit of normal (ULN).
6. History of HIV-2, hepatitis B and/or C, cirrhosis of the liver, or any known active or chronic liver disease. Hepatitis B vaccinated patients are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To determine the percentage of patients who achieve HIV-1 RNA levels below 50 copies/mL at Week 24 | 24 weeks

CONTACTS AND LOCATIONS:
Locations (48):
- United States (45):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Southwest Center for HIV / AIDS, Phoenix, Arizona
  - AIDS Healthcare Foundation Research Center, Beverly Hills, California
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Providence Clinical Research, Burbank, California
  - AIDS Research Alliance, Los Angeles, California
  - Peter J Ruane MD Incorporated, Los Angeles, California
  - Oasis Clinic, Los Angeles, California
  - Anthony Mills, Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - Stanford University ACTU, Palo Alto, California
  - University of California at San Francisco, San Francisco, California
  - Quest Clinical Research, San Francisco, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Whitman-Walker Clinic, Washington D.C., District of Columbia
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Gary Richmond, Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Care Resource Inc., Miami, Florida
  - Kinder Medical Group, Miami, Florida
  - Wohlfeiler, Piperato & Associates, LLC, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Health Positive, Safety Harbor, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - Triple O Research Institute, PA, West Palm Beach, Florida
  - AIDS Research Consortium of Atlanta, Inc., Atlanta, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - Community Research Initiative of New England, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - ID Care, Hillsborough, New Jersey
  - Synergy First Medical PLLC, Brooklyn, New York
  - Erie County Medical Center Corporation, Buffalo, New York
  - Bisher Akil, M.D., A Medical Corporation, New York, New York
  - Aaron Diamond AIDS Research Center, New York, New York
  - ACRIA, New York, New York
  - Jacobi Medical Center, New York, New York
  - AIDS Care, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Rosedale Infectious Disease, Huntersville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - North Texas Infectious Diesease Consultants, Dallas, Texas
  - Therapeutic Concepts, Houston, Texas
  - The University of Texas Health Science Center at Houston Medical School, Houston, Texas
- Puerto Rico (3):
  - Univ. of Puerto Rico - ACTU, San Juan, PR
  - University of Puerto Rico, School of Medicine, CEMI, San Juan, PR
  - Clinical Research P.R., Inc., Santurce, Puerto Rico

REFERENCES:
- [Derived] Sherman KE, Abdel-Hameed E, Rouster SD, Shata MTM, Blackard JT, Safaie P, Kroner B, Preiss L, Horn PS, Kottilil S. Improvement in Hepatic Fibrosis Biomarkers Associated With Chemokine Receptor Inactivation Through Mutation or Therapeutic Blockade. Clin Infect Dis. 2019 May 17;68(11):1911-1918. doi: 10.1093/cid/ciy807. PMID 30239650
- [Derived] Thompson M, Saag M, DeJesus E, Gathe J, Lalezari J, Landay AL, Cade J, Enejosa J, Lefebvre E, Feinberg J. A 48-week randomized phase 2b study evaluating cenicriviroc versus efavirenz in treatment-naive HIV-infected adults with C-C chemokine receptor type 5-tropic virus. AIDS. 2016 Mar 27;30(6):869-78. doi: 10.1097/QAD.0000000000000988. PMID 26636929
- [Derived] Kagan RM, Johnson EP, Siaw MF, Van Baelen B, Ogden R, Platt JL, Pesano RL, Lefebvre E. Comparison of genotypic and phenotypic HIV type 1 tropism assay: results from the screening samples of Cenicriviroc Study 202, a randomized phase II trial in treatment-naive subjects. AIDS Res Hum Retroviruses. 2014 Feb;30(2):151-9. doi: 10.1089/AID.2013.0123. Epub 2013 Aug 14. PMID 23875707